CLINICAL TRIAL: NCT00002307
Title: A Double-Blind Comparison of Zidovudine (AZT) Versus Stavudine (d4T; BMY 27857) for the Treatment of Patients With HIV Infection Who Have Absolute CD4 Lymphocyte Counts Between 50 and 500 Cells/mm3
Brief Title: A Comparison of Zidovudine (AZT) and Stavudine in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 116A; AI455-019
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: HIV Infections
Keywords: Zidovudine; Stavudine
MeSH Terms: conditions — HIV Infections | interventions — Stavudine; Zidovudine

INTERVENTIONS:
Drug: Stavudine
Drug: Zidovudine

SUMMARY:
To compare stavudine (d4T) and zidovudine (AZT) in slowing the progression of HIV disease. To compare the antiviral activity of d4T versus AZT as measured by plasma levels of p24 antigen and HIV viremia, and their relative efficacy by improvement and/or absence of adverse changes over time in laboratory parameters associated with HIV infection. To compare the safety of oral doses of d4T to AZT in patients with HIV infection.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* AZT.

Patients must have:

* Documented HIV infection as determined by a positive ELISA and/or Western blot.
* Absolute CD4 count of 100 - 500 cells/mm3 within 90 days prior to registration OR a CD4 count of 50 - 99 cells/mm3 within 30 days prior to registration.
* Prior zidovudine therapy for at least 6 months and currently tolerating at least 500 mg daily.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Newly diagnosed AIDS-defining opportunistic infection requiring acute therapy at time of enrollment.
* Need for chronic systemic therapy at time of enrollment.
* Intractable diarrhea.
* Signs or symptoms of bilateral peripheral neuropathy at time of screening.
* Demonstrated intolerance to zidovudine therapy.
* Any other clinical conditions that would render the patient unsuitable for study or unable to comply with the dosing requirements.

Concurrent Medication:

Excluded:

* Chronic systemic therapy with agents likely to suppress bone marrow, cause neurotoxicity, or create hepatic dysfunction.

Patients with the following prior conditions are excluded:

* Prior history of bilateral peripheral neuropathy.
* Demonstrated intolerance to zidovudine therapy.

Prior Medication:

Excluded:

* Prior d4T, ddI, or ddC.
* Other investigational antiretroviral drugs (e.g., AZddU, Al 721, interferon, or immunomodulating drugs within 1 month prior to study entry or ribavirin within 3 months prior to study entry).
* Prior myelosuppressive, neurotoxic, or cytotoxic anticancer therapy within 3 months prior to study entry.
* Any prior therapy that would render the patient unsuitable for study or unable to comply with dosing requirements.

Required:

* At least 6 months of prior AZT and currently tolerating at least 500 mg daily, with the last dose received no more than 7 days prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Study Completion 1994-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (44):
  - Univ of Arizona / Health Science Ctr, Tucson, Arizona
  - East Bay AIDS Ctr, Berkeley, California
  - Children's Hosp of Los Angeles, Los Angeles, California
  - Combat Group, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Cedars Sinai Med Ctr, Los Angeles, California
  - UCD Med Ctr / AIDS and Related Disorders Clinic, Sacramento, California
  - Children's Hosp of San Francisco, San Francisco, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Whitman - Walker Clinic, Washington D.C., District of Columbia
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Community Research Initiative of South Florida, Coral Gables, Florida
  - TheraFirst Med Ctrs Inc, Fort Lauderdale, Florida
  - Univ of Miami, Miami, Florida
  - Infectious Disease Research Institute Inc, Tampa, Florida
  - Dr Steven Marlowe, Atlanta, Georgia
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Infectious Diseases Research Clinic / Indiana Univ Hosp, Indianapolis, Indiana
  - Univ of Kansas School of Medicine / Univ Hosp, Kansas City, Kansas
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Chase Braxton Health Service, Baltimore, Maryland
  - New England Deaconess Hosp, Boston, Massachusetts
  - Univ of Nebraska Med Ctr / HIV Clinic, Omaha, Nebraska
  - Univ of New Mexico School of Medicine, Albuquerque, New Mexico
  - Beth Israel Med Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Cornell Univ Med College, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - SUNY / Health Sciences Ctr at Stony Brook, Stony Brook, New York
  - Bronx Veterans Affairs Med Ctr, The Bronx, New York
  - Nalle Clinic, Charlotte, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Pennsylvania / HIV Clinic, Philadelphia, Pennsylvania
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Montefiore Hosp, Pittsburgh, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Dr Edward Stool, Houston, Texas
  - Houston Clinical Research Network, Houston, Texas
  - Univ TX San Antonio Health Science Ctr, San Antonio, Texas
  - Univ of Utah School of Medicine, Salt Lake City, Utah
  - Milwaukee County Med Complex, Milwaukee, Wisconsin
- UPR School of Medicine / San Juan Veterans Adm Med Ctr, San Juan, Puerto Rico

REFERENCES:
- [Background] Spruance SL, Pavia AT, Mellors JW, Murphy R, Gathe J Jr, Stool E, Jemsek JG, Dellamonica P, Cross A, Dunkle L. Clinical efficacy of monotherapy with stavudine compared with zidovudine in HIV-infected, zidovudine-experienced patients. A randomized, double-blind, controlled trial. Bristol-Myers Squibb Stavudine/019 Study Group. Ann Intern Med. 1997 Mar 1;126(5):355-63. doi: 10.7326/0003-4819-126-5-199703010-00003. PMID 9054279